CLINICAL TRIAL: NCT01097447
Title: Collagen Crosslinking With Ultraviolet-A in Asymmetric Corneas
Brief Title: Collagen Crosslinking With Ultraviolet-A in Asymmetric Corneas (2)
Status: Terminated | Type: Observational
Why Stopped: Terminated to initiate FDA IND-cleared study protocol
Sponsor: Cxlusa (Industry)
Responsible Party: Sponsor
Other Study IDs: CXL (2)
Record Dates: First submitted 2010-03-25; First posted 2010-04-01 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Keratoconus; Ectasia; Degeneration
Keywords: Diagnosis of keratoconus, post-LASIK ectasia, FFKC, or pellucid marginal degeneration
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ciprofloxicine or Vigamox or other: up to qid till epithelialized.
- Topical Nonsteroidal (Acular, Acuvail, Voltaren Xibrom: up to qid for up to 5-10 days postop
- Topical steroid (FML, Pred Forte, Flarex: qid for up to 8 weeks

SUMMARY:
To evaluate the efficacy of ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) as a method to increase the biomechanical and biochemical stability of the cornea by inducing additional cross-links within or between collagen fibers using UVA light and the photo- mediator riboflavin. The purpose of this study is to generate data for presentation at medical meetings and for peer-review publication

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age or older
* Diagnosis of keratoconus, post-LASIK ectasia, or pellucid marginal degeneration or forme fruste pellucid marginal degeneration.
* Diagnosis of FFKC
* History of Radial Keratotomy with fluctuating vision.
* Ability to provide written informed consent
* Likely to complete all study visits
* Minimum corneal thickness of at least 300 measured by ultrasound or Pentacam

Exclusion Criteria:

* Severe corneal scarring that markedly affects vision
* Contraindications to any study medications or their components
* Pregnancy or breast feeding
* Active Herpes Corneal Disease

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 2619 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Increase the biomechanical and biochemical stability of the cornea by inducing additional cross-links within | 1 year

SECONDARY OUTCOMES:
increase the biomechanical and biochemical stability of the cornea between collagen fibers using UVA light and the photo- mediator riboflavin | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Parag Majmudar, MD, Principal Investigator — Chicago Cornea Consultants, LTD; Lance Forstot, MD, Principal Investigator — Corneal Consultants of Colorado, P.C; Bradley Bowman, M.D, Principal Investigator — Cornea Associates of Texas; Sandy Feldman, M.D, Principal Investigator — Clear View Eye & Laser Medical Center; Sherman Reeves, MD, Principal Investigator — Minnesota Eye Consultants, P.A.
Locations (5):
- United States (5):
  - Clear View Eye & Laser Medical Center, San Diego, California
  - Corneal Consultants of Colorado, P.C, Littleton, Colorado
  - Chicago Cornea Consultants, LTD, Hoffman Estates, Illinois
  - Minnesota Eye Consultants, P.A., Bloomington, Minnesota
  - Cornea Associates of Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No